CLINICAL TRIAL: NCT04217668
Title: Pain Perception, Headache Provocation and Multiomics of People Who Are Unable to Have Headache
Brief Title: Headache Provocation of People Who Are Unable to Have Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Isa Amalie Olofsson, Medical Doctor, PhD student, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HR002 Provocation
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Headache; Healthy
MeSH Terms: conditions — Headache | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Intervention Model Description: Blinded case-control study
Masking Description: The investigators are blinded to the case-control grouping of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isosorbide mononitrate (Experimental): Cases and controls both receive one tablet Imdur® 60 mg (isosorbide mononitrate) on the study day.
  Interventions: Drug: Isosorbide Mononitrate 60 MG

INTERVENTIONS:
Drug: Isosorbide Mononitrate 60 MG — 1 tablet Isosorbide Mononitrate 60 mg administrated orally.
  Other Names: Imdur

SUMMARY:
Headaches are extremely common illnesses with a combined lifetime prevalence of 90-99% in Europe. Despite this high prevalence, there are persons who have never, in their whole life, encountered a headache.

The aim of the study is to identify factors that protect against headache by studying headache after provocation in people who never have had a headache (headache resistant) versus non-resistant controls.

The investigators will use isosorbide mononitrate as a pharmacological trigger of headache. The provocation is performed by investigators who are blinded to the grouping of the participants.

The investigators hope to contribute with novelty to the current understanding of headache pathophysiology and development of more efficient treatment of headache.

ELIGIBILITY:
Inclusion Criteria:

* Headache resistant and non-resistant male participants from the Danish Blood Donor Study.
* Weight: 45 kg to 95 kg

Exclusion Criteria:

* Daily consumption of any medication.
* Consumption of any medication less than 12 hours prior to the study day.
* Headache on the study day or 48 hours prior to the study day.
* Amnestic or clinical signs of hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) or hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg).
* Any severe cardiovascular disease, including cerebrovascular illness.
* Amnestic or clinical signs of current mental illness.
* Amnestic or clinical signs of current substance or drug abuse.
* Amnestic or clinical signs of any illness the responsible doctor considers relevant for participation in the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve of headache intensity | 5 hours
  Area under the curve of headache intensity from 0 - 5 hours post tablet administration

SECONDARY OUTCOMES:
Area under the curve of headache intensity | 12 hours
  Area under the curve of headache intensity from 0 - 12 hours post tablet administration

CONTACTS AND LOCATIONS:
Overall Officials: Jes Olesen, Professor, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Region H, Denmark

IPD SHARING:
Plan to Share IPD: Undecided